CLINICAL TRIAL: NCT04342208
Title: Evaluate the Working Environments of Individuals Working From Home During Covid-19 Outbreak
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Polen Akşimşek, PhD student, Istanbul University - Cerrahpasa
Other Study IDs: GPA1347
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the working environments of individuals working from home during the covid-19 outbreak and the effect of the working environments on their musculoskeletal system.

DETAILED DESCRIPTION:
The study will include people between the ages of 18-65 who work from home (works in the office before isolation) as a part of the Covid-19 isolation measure. The working environment of the individuals participating in the study will be evaluated with The Rapid Office Strain Assessment (ROSA). Musculoskeletal symptoms will be analyzed by using the Standardised Nordic Questionnaires (NMQ). Pain will be analyzed by using the Visual Analogue Scale (VAS) .

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* works from home
* works in the office before isolation

Exclusion Criteria:

* have any systemic disease that may affect on musculoskeletal system such as fibromyalgia, myofacial pain syndrome, etc.
* have any vision problem
* have difficulty of understanding and following online survey
* have any physical disability
* have self-reported computer use for less than four hours on a typical workday

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include people between the ages of 18-65 who works from home (works in the office before isolation) as a part of Covid-19 isolation measure
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
The Rapid Office Strain Assessment (ROSA) | 30 minutes
  The working environment of the individuals participating in the study will be evaluated with The Rapid Office Strain Assessment (ROSA). ROSA is a picture-based posture checklist designed to quantify exposure to risk factors in an office work environment. In ROSA, three subsections (A-chair height, depth, armrest, and backrest; B-monitor and telephone; C-mouse and keyboard) of the office work environment are assessed. After completing the ROSA checklist, the related tables are used to calculate the score from each part, and eventually, the final ROSA score is derived. If the final score is ≤4; the risk of musculoskeletal disorders is low (low risky). If the final score is ≥5 the risk of musculoskeletal disorders risk is high (high risky).

SECONDARY OUTCOMES:
The Standardised Nordic Questionnaries (NMQ) | 15 minutes
  The NMQ includes 27 items exploring the presence of musculoskeletal symptoms for the last 12 months covering nine different parts of the body. It also has items about severity grades, determined according to functional status and the presence of musculoskeletal symptoms during the 7 days. Symptoms indicate musculoskeletal disorders in different body regions among the working population. The NMQ section that questions the last 7 days will be used in the study. In that section consists additional questions relating to the neck, the shoulders, and the lower back further detail relevant issues. Twenty-five forced-choice questions elicit any accidents affecting each area, functional impact at home and work (change of job or duties), duration of the problem, assessment by a health professional, and musculoskeletal problems in the last 7 days.

OTHER OUTCOMES:
Visual Analog Scale (VAS) | 2 minutes
  Pain will be analyzed by using the Visual Analogue Scale (VAS). VAS is a scale assessing pain intensity and composed of a horizontal or vertical line and anchored at both ends by words indicative of extremes of magnitude, such as "no pain" to "most intense pain sensation imaginable". In the current study, at the last 1 year and last 7 days, pain intensity was assessed by using horizontal lined VAS. Higher values show higher pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barbieri DF, Srinivasan D, Mathiassen SE, Oliveira AB. Variation in upper extremity, neck and trunk postures when performing computer work at a sit-stand station. Appl Ergon. 2019 Feb;75:120-128. doi: 10.1016/j.apergo.2018.09.012. Epub 2018 Oct 3. PMID 30509516
- [Background] Brewer S, Van Eerd D, Amick BC 3rd, Irvin E, Daum KM, Gerr F, Moore JS, Cullen K, Rempel D. Workplace interventions to prevent musculoskeletal and visual symptoms and disorders among computer users: a systematic review. J Occup Rehabil. 2006 Sep;16(3):325-58. doi: 10.1007/s10926-006-9031-6. PMID 16933148
- [Background] Sonne M, Villalta DL, Andrews DM. Development and evaluation of an office ergonomic risk checklist: ROSA--rapid office strain assessment. Appl Ergon. 2012 Jan;43(1):98-108. doi: 10.1016/j.apergo.2011.03.008. Epub 2011 May 6. PMID 21529772
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Clark P, Lavielle P, Martinez H. Learning from pain scales: patient perspective. J Rheumatol. 2003 Jul;30(7):1584-8. PMID 12858463
- [Background] Kahraman T, Genc A, Goz E. The Nordic Musculoskeletal Questionnaire: cross-cultural adaptation into Turkish assessing its psychometric properties. Disabil Rehabil. 2016 Oct;38(21):2153-60. doi: 10.3109/09638288.2015.1114034. Epub 2016 Jan 4. PMID 26726840
- See also: Related Info — http://www.apta.org/uploadedFiles/APTAorg/News_and_Publications/Latest_News/News_Items/2020/Physiotherapy_Guideline_COVID-19.pdf
- See also: Related Info — http://www.who.int/emergencies/diseases/novel-coronavirus-2019/advice-for-public